CLINICAL TRIAL: NCT02348554
Title: A Smartphone Application to Evaluate Energy Expenditure and Duration of Activities in Free-living Conditions for Overweight and Obese People (eMouve3)
Brief Title: A Smartphone Application to Evaluate Energy Expenditure and Duration of Activities for Overweight and Obese People
Acronym: eMouve3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Almerys (Other)
Responsible Party: Principal Investigator, Martine DUCLOS, Physician, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AU1070; 2013-A01140-45 (Other: ANSM)
Record Dates: First submitted 2014-09-26; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Obesity; Physical Activity
Keywords: obesity; energy expenditure; daily living physical activity; smartphone; accelerometry; prediction algorithm
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Controlled conditions (Experimental): Volunteers were asked to perform several activities such as walking at different paces, running, sitting, standing still or taking public transportation for about 1h30 They wore 3 research sensors that estimated energy expenditure: Fitmate, Armband and Actiheart. They also wore smartphones (in front pant pockets) that collected accelerometry data.
  Interventions: Behavioral: Controlled conditions
- Free-living conditions (Experimental): Volunteers were asked to wear sensors during about 12 hours, one day. They wore 2 research sensors that estimated energy expenditure: Armband and Actiheart. They also wore smartphones (in front pant pockets) that collected accelerometry data.
  Interventions: Behavioral: Free-living conditions

INTERVENTIONS:
Behavioral: Controlled conditions — The 13 volunteers in controlled conditions performed each of the nine activities several times according to the activity scenario: sitting, slow, normal and brisk walking, climbing and descending stairs (eight floors), standing, slow running and taking public transportation (tramway). The duration of each activity varied from 2 to 20 minutes.
  Arms: Controlled conditions
Behavioral: Free-living conditions — The spontaneous activities of 30 volunteers were recorded in the free-living conditions for a full day selected either during the week or the weekend.
  Arms: Free-living conditions

SUMMARY:
The aim of this study was to validate functions for estimating energy expenditure in controlled and free-living conditions. This method was based on accelerometry data acquired from smartphones worn in a trouser pocket. The developed functions have been compared to the estimations provided by three research devices named Fitmate, Armband and Actiheart.

DETAILED DESCRIPTION:
There is a growing interest in evaluating physical activity and energy expenditure (EE) to provide feedback to the user. The use of mass-market sensors such as accelerometers offers a promising solution for the general public due to the growing smartphone market over the last decade.

Two previous studies allowed to propose a function named PredEE, which has been tested on normal-weighted volunteers.

This EE estimation function has been tested and improved with data collected from 43 overweight volunteers equipped with smartphones and two or three research sensors (Fitmate, Armband and Actiheart in controlled conditions, and Armband and Actiheart in free-living conditions). Research sensors' data serves as reference during the evaluation and improvement of the proposed function.

This EE estimation function using the smartphone technology is dedicated to light- and moderate-intensity activities, and the investigators believe it can be a new way to help people controlling their daily physical activity level.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* age: 18-60 years
* BMI between 28 and 42 kg/m²
* subject considered as healthy after clinical examination and medical questionnaire
* no pregnant women
* subject with normal rest electrocardiogram (validated by a cardiologist)
* certificate of non-indication against the practice of exercise stress testing delivered by a physician
* subject with normal blood pressure (<140/90 mm Hg) with or without medical treatment
* subject with no foot pad problem
* subject giving his/her written informed consent
* subject willing to comply with study procedures
* affiliated to National Health Insurance

Exclusion Criteria:

* respiratory failure or cardiovascular problem
* non-indication against the practice of exercise stress testing
* known cardiac decompensation or myocardial infarction
* surgery made less than 6 months before the study beginning
* pregnant women and nursing mother
* current infectious pathology
* abnormal electrocardiogram
* not affiliated to national health insurance people
* under legal guardianship
* refusal to sign informed consent
* refusal to be registered on the national volunteers data file
* currently participating or who having got 4500€ in this year before to have participated in another clinical trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Accelerometry | 1 day
  Measures acquired by smartphones including a tri-axial accelerometer

SECONDARY OUTCOMES:
Energy expenditure | 1 day
  Sensor: Fitmate
Energy expenditure | 1 day
  Sensor: Armband
Energy expenditure | 1 day
  Sensor: Actiheart

OTHER OUTCOMES:
Rest energy expenditure | 1 day
  Measurement of rest energy expenditure under canopy by Fitmate
Rest energy expenditure | 1 day
  Measurement of rest energy expenditure by using Armband
Rest energy expenditure | 1 day
  Measurement of rest energy expenditure by using Actiheart

CONTACTS AND LOCATIONS:
Overall Officials: Martine Duclos, Physician, Principal Investigator — CHU G Montpied
Locations (1):
- Centre de Recherche en Nutrition Humaine d'Auvergne, Clermont-Ferrand, France

REFERENCES:
- [Background] Rousset S, Fardet A, Lacomme P, Normand S, Montaurier C, Boirie Y, Morio B. Comparison of total energy expenditure assessed by two devices in controlled and free-living conditions. Eur J Sport Sci. 2015;15(5):391-9. doi: 10.1080/17461391.2014.949309. Epub 2014 Aug 21. PMID 25141769
- [Background] Guidoux R, Duclos M, Fleury G, Lacomme P, Lamaudiere N, Manenq PH, Paris L, Ren L, Rousset S. A smartphone-driven methodology for estimating physical activities and energy expenditure in free living conditions. J Biomed Inform. 2014 Dec;52:271-8. doi: 10.1016/j.jbi.2014.07.009. Epub 2014 Jul 15. PMID 25048352
- See also: the site ActivCollector collects and processes accelerometry data sent by the smartphones, and then ActivCollector sends the EE and activity durations results to the smartphone's user — http://activcollector.clermont.inra.fr/home